CLINICAL TRIAL: NCT04177225
Title: Evaluation of Dynamic Monitors for the Prediction of Volume Responsiveness in Patients With and Without Diastolic Dysfunction
Brief Title: Effect of Diastolic Dysfunction on Dynamic Cardiac Monitors
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1380344
Record Dates: First submitted 2019-04-19; First posted 2019-11-26 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Stroke Volume Variation; Diastolic Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with normal diastolic function: Patients undergoing scheduled surgical procedures requiring general anesthesia and invasive arterial pressure and advanced cardiac function monitoring. A trans thoracic ultrasound examination of cardiac function will be performed before induction of general anesthesia . In the operating room, the anesthesia care team will place all of the standard intra-operative monitors and then induce general anesthesia. After induction, the ultrasound examination will be repeated and the planned additional intra-operative monitors will be placed. The arterial catheter will be attached to a FloTrac/EV1000 monitor that will be used to guide fluid management during the procedure. The sensitivity and specificity of SVV to predict the response of cardiac output to intravenous fluid administration will be assessed in this patient group distinguished by their normal left ventricular diastolic function.
  Interventions: Procedure: Trans thoracic Ultrasound Examination; Other: Intravenous fluid administration
- Patients with abnormal diastolic function: Patients undergoing scheduled surgical procedures requiring general anesthesia and invasive arterial pressure and advanced cardiac function monitoring. A trans thoracic ultrasound examination of cardiac function will be performed before induction of general anesthesia . In the operating room, the anesthesia care team will place all of the standard intra-operative monitors and then induce general anesthesia. After induction, the ultrasound examination will be repeated and the planned additional intra-operative monitors will be placed. The arterial catheter will be attached to a FloTrac/EV1000 monitor that will be used to guide fluid management during the procedure. The sensitivity and specificity of SVV to predict the response of cardiac output to intravenous fluid administration will be assessed in this patient group distinguished by their abnormal left ventricular diastolic function.
  Interventions: Procedure: Trans thoracic Ultrasound Examination; Other: Intravenous fluid administration

INTERVENTIONS:
Procedure: Trans thoracic Ultrasound Examination — Ultrasound examination of cardiac function before and after induction of general anesthesia.
Other: Intravenous fluid administration — Intravenous fluids will be administered as a bolus in response to standard clinical indications

SUMMARY:
This investigator initiated, prospective, observational, single-center study is designed to assess whether dynamic monitors of cardiac function such as stroke volume variation (SVV) that have been shown to predict volume responsiveness differ in clinical utility between patients with and without diastolic dysfunction.

DETAILED DESCRIPTION:
This investigator initiated, prospective, observational, single-center study is designed to assess whether dynamic monitors of cardiac function, such as stroke volume variation (SVV), that have been shown to predict volume responsiveness differ in clinical utility between patients with and without diastolic dysfunction.

Specific Aims:

* Determine the threshold for the predictive response of SVV with respect to increasing cardiac output for patients with and without diastolic dysfunction.
* Compare the trans thoracic ultrasound assessment of left ventricular diastolic function before and after the induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients Undergoing Elective surgical procedures where invasive arterial line pressure monitoring is a planned part of the intraoperative management
* Age greater than or equal to 18
* Procedures requiring general anesthesia and mechanical ventilation

Exclusion Criteria:

* Adults unable to provide consent
* Atrial Fibrillation or other significant active arrhythmia
* Emergency Procedures
* Hemodynamic instability requiring vasopressor and/or inotropic infusions
* Presence of an intra-aortic balloon pump
* Open thoracic procedures
* Extremes of BMI less than 20 or greater than 40
* Pregnancy
* Prisoners
* Patient Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgical procedures requiring arterial line pressure monitoring at the University of California Davis Medical Center Surgical Unit
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Impact of diastolic function on the response threshold for stroke volume variation (SVV) as a predictor of the cardiac output response to fluid administration. | Through study completion, an average of 1 year
  The sensitivity of SVV as a predictor of the change in cardiac output in response to IV fluid administration will be determined by analysis of the Receiver Operator Characteristic (ROC) curves for each of the patient groups as distinguished by their pre-induction assessment of diastolic left ventricular function

SECONDARY OUTCOMES:
Grade assessment of diastolic function | Through study completion, an average of 1 year
  Transthoracic ultrasound will be performed before and after the induction of general anesthesia to assess left ventricular diastolic function. Measurements of trans-mitral flow velocities and tissue Doppler velocities will be used to establish the grade of left ventricular diastolic function. The reproducibility of this measurement before and after the induction of anesthesia has ramifications for intra-operative measurement of diastolic function.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Fleming, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Health System, Sacramento, California, United States

REFERENCES:
- [Derived] Desai S, Hamilton Z, McCloskey L, Badakhsh O, Li D, Fleming NW. The effect of propofol on the grading of diastolic function: a prospective observational study. BMC Anesthesiol. 2025 Jul 30;25(1):376. doi: 10.1186/s12871-025-03260-2. PMID 40739534
- [Derived] Abdallah AC, Song SH, Fleming NW. A retrospective study of the effects of a vasopressor bolus on systolic slope (dP/dt) and dynamic arterial elastance (Eadyn). BMC Anesthesiol. 2024 Jul 29;24(1):257. doi: 10.1186/s12871-024-02574-x. PMID 39075354